CLINICAL TRIAL: NCT04419545
Title: Covid Radiographic Images Data-set for A.I
Acronym: CORDA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: University of Turin, Italy (Other); Azienda Ospedaliera Ordine Mauriziano di Torino (Other)
Responsible Party: Principal Investigator, Giorgio Limerutti, M.D., A.O.U. Città della Salute e della Scienza
Other Study IDs: CORDA
Record Dates: First submitted 2020-06-04; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Radiology; Artificial Intelligence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- interstitial pneumonia cases: Chest x-ray diagnosis
  Interventions: Diagnostic Test: Neural network diagnosis algorithm
- Negative controls: Chest x-ray Negative for pneumonia
  Interventions: Diagnostic Test: Neural network diagnosis algorithm

INTERVENTIONS:
Diagnostic Test: Neural network diagnosis algorithm — we feed neural network with chest x-ray radiography images for teaching the network for automatic diagnosis of interstitial pneumonia

SUMMARY:
The possibility to use widespread and simple chest X-ray (CXR) imaging for early screening of COVID-19 patients is attracting much interest from both the clinical and the Artificial intelligence community. In this study we provide insights and also raise warnings on what is reasonable to expect by applying deep learning to COVID classification of CXR images. We provide a methodological guide and critical reading of an extensive set of statistical results that can be obtained using currently available datasets. In particular, we take the challenge posed by current small size COVID data and show how significant can be the bias introduced by transfer-learning using larger public non- COVID CXR datasets. We also contribute by providing results on a medium size COVID CXR dataset, just collected by one of the major emergency hospitals in Northern Italy during the peak of the COVID pandemic. These novel data allow us to contribute to validate the generalization capacity of preliminary results circulating in the scientific community. Our conclusions shed some light into the possibility to effectively discriminate COVID using CXR.

DETAILED DESCRIPTION:
COVID-19 virus has rapidly spread in mainland China and into multiple countries worldwide. As of April 7th 2020 in Italy, one of the most severely affected countries, 135,586 Patients with COVID19 were recorded, and 17,127 of them died; at the time of writing Piedmont is the 3rd most affected region in Italy, with 13,343 recorded cases. Early diagnosis is a key element for proper treatment of the patients and prevention of the spread of the disease. Given the high tropism of COVID-19 for respiratory airways and lung epithelium, identification of lung involvement in infected patients can be relevant for treatment and monitoring of the disease. Virus testing is currently considered the only specific method of diagnosis. The Center for Disease Control (CDC) in the US recommends collecting and testing specimens from the upper respiratory tract (nasopharyngeal and oropharyngeal swabs) or from the lower respiratory tract when available (bronchoalveolar lavage, BAL) for viral testing with reverse transcription polymerase chain reaction (RT-PCR) assay. Current position papers from radiological societies (Fleischner Society, SIRM, RSNA) do not recommend routine use of imaging for COVID-19 diagnosis.

However, it has been widely demonstrated that, even at early stages of the disease, chest x-rays (CXR) and computed tomography (CT) scans can show pathological findings. It should be noted that they are actually non specific, and overlap with other viral infections (such as influenza, H1N1, SARS and MERS): most authors report peripheral bilateral ill-defined and ground-glass opacities, mainly involving the lower lobes, progressively increasing in extension as disease becomes more severe and leading to diffuse parenchymal consolidation, CT is a sensitive tool for early detection of peripheral ground glass opacities; however routine role of CT imaging in these Patients is logistically challenging in terms of safety for health professionals and other patients, and can overwhelm available resources. Chest X-ray can be a useful tool, especially in emergency settings: it can help exclude other possible lung "noxa", allow a first rough valuation of the extent of lung involvement and most importantly can be obtained at patients bed using portable devices, limiting possible exposure in health care workers and other patients. Furthermore, CXR can be repeated over time to monitor the evolution of lung disease.

Methodology:

we describe the deeplearning approach based on quite standard pipeline, namely chest image pre-processing and lung segmentation followed by classification model obtained with transfer learning. As we will see in this section, data pre-processing is fundamental to remove any bias present in the data. In particular, we will show that it is easy for a deep model to recognize these biases which drive the learning process. Given the small size of COVID datasets, a key role is played by the larger datasets used for pre-training. Therefore, we first discuss which datasets can be used for our goals.

ELIGIBILITY:
Inclusion Criteria: chest x ray performed during emergency department or hospital stay

-

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the people treated in radiology dept
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
sensibility and specificity of neural network diagnosis | at day 0
  sensibility and specificity of neural network diagnosis compared with human diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Limerutti, M.D., Principal Investigator — Radiology Unit A.O.U. Città della Salute e della Scienza
Locations (1):
- Azienda Ospedaliero Universitaria Città della Salute e della Scienza, Torino, Turin, Italy

IPD SHARING:
Plan to Share IPD: No